CLINICAL TRIAL: NCT03896815
Title: Expanded Access Use of INCB054329 to Treat a Single Patient With Metastatic Renal Cell Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-54329-17-01
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

MeSH Terms: interventions — INCB054329

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: INCB054329

SUMMARY:
Expanded access use of INCB054329 to treat a single patient with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Schneider, MD, Principal Investigator — University of Michigan